CLINICAL TRIAL: NCT07175363
Title: The Application of Butorphanol in Postoperative Analgesia Management After Cesarean Section: A Retrospective Cohort Study
Brief Title: Butorphanol for Pain Relief After Cesarean Section: A Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yanyu Liu, Physician-in-charge, Sichuan Provincial People's Hospital
Other Study IDs: 2025-598
Record Dates: First submitted 2025-09-07; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Caesarean Section
Keywords: Caesarean section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The group using the analgesic pump
  Interventions: Drug: An postoperative analgesic pump was used

INTERVENTIONS:
Drug: An postoperative analgesic pump was used — The drugs in the analgesic pump include butorphanol, hydromorphone, tramadol, and other medications.

SUMMARY:
This study explored the association between postoperative functional recovery and the formula of analgesic pumps as well as other related factors (such as age, intraoperative blood loss, operation duration, etc.) by retrospectively analyzing the clinical data of patients undergoing cesarean section in the main campus and branches of Sichuan Provincial People's Hospital from September 2024 to June 2025. The value of this study lies in: 1) providing a basis for optimizing the postoperative analgesia plan after cesarean section. 2) To provide references for the formulation of personalized analgesia strategies in clinical practice, improve the postoperative recovery quality of patients, promote the concept of enhanced recovery after surgery, and reduce the medical burden.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 years
2. ASAI-III level
3. Scheduled or emergency cesarean section
4. Postoperative use of analgesic pump (formulation includes buprenorphine or tramadol or hydromorphone, etc.)
5. Complete electronic medical records

Exclusion Criteria:

1. Postoperative analgesia pump usage time is less than 24 hours
2. Missing key information such as follow-up status in medical records

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who have given birth by cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 2 days post-surgery
  The Visual Analog Scale (VAS) is primarily used, where 1 represents no pain (best outcome) and 10 represents the worst pain (worst outcome); other scales may be used if necessary.
Postoperative functional recovery status | 2 days post-surgery
  Postoperative functional recovery status mainly includes: the time of first passage of gas, the time of first ambulation, the time of first catheter removal, and the recovery of limb muscle strength. The passage of gas, ambulation, and catheter removal times are self-reported by the patients, recording the days after surgery when the events occurred. The recovery of limb muscle strength is classified into six levels, ranging from 0 to 5, where 0 indicates no detectable muscle contraction (worst outcome) and 5 indicates normal muscle strength (best outcome).
Sedation score | 2 days post-surgery
  The sedation score uses a scale from -5 to +4, where -5 is defined as coma (one of the worst outcomes); -4 is defined as severe sedation (responds to physical stimulation); -3 is moderate sedation (no response to auditory stimulation); -2 is mild sedation (unable to maintain alertness for more than 10 seconds); -1 is drowsiness (not fully awake but can stay awake for more than 10 seconds); 0 is the awake natural state (best outcome); +1 is restlessness and anxiety (anxious and tense, but only slight body movement); +2 is agitation and anxiety (intense body movement); +3 is very agitated (trying to remove body tubes); +4 is aggressive (violent behavior) (one of the worst outcomes).

SECONDARY OUTCOMES:
Overall patient satisfaction rating | 2 days post-surgery
  Patient overall satisfaction is self-reported, with a score range from 0 to 100, where 0 represents the least satisfied (worst outcome) and 100 represents the most satisfied (best outcome).
Nausea and vomiting | 2 days post-surgery
  Self-reported by the patient, with '1' indicating occurrence (worst outcome) and '0' indicating non-occurrence (best outcome).
Adverse reactions | 2 days post-surgery

IPD SHARING:
Plan to Share IPD: No